CLINICAL TRIAL: NCT05780398
Title: Long Term Follow up in Pediatric Supracondylar Humeral Fracture After Surgical Treatment
Brief Title: Long Term Follow up in Pediatric Supracondylar Humeral Fracture
Acronym: SUPCONFOLLOW
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0384
Record Dates: First submitted 2023-03-04; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Supracondylar Humerus Fracture; Elbow Fracture
Keywords: long term follow up
MeSH Terms: conditions — Elbow Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to learn about long term outcomes in Supracondylar Humeral Fracture in children after surgery.

The main questions it aims to answer are:

* how good is the elbow function
* what are the post-operative complication
* what is the time before return to sport
* what is the aesthetic prejudice of the scar for the patient Participants will answer questionnaries and send photographs of their elbows to the examinator

DETAILED DESCRIPTION:
Elbow fractures represent 5% of total fracture in children. Supracondylar humeral fractures compound half of them.

As distal humerus is responsible for only 20% of humeral growth, bone remodelage her is less important compared to other sites in children..

Many different attitudes are possible : orthopedic reduction, open reduction, percutaneous pinning ... No methode as clearly demontrated a superiority.

Percutaneous pinning as been widely used the last years though We haven't find any study evaluating long term outcomes regarding functionnal and aesthetic outcomes in supracondylar humeral fracture treated by percutaneous pinning.

ELIGIBILITY:
Inclusion Criteria:

* Children operated for a supracondylar humeral fracture in university hospital of Grenoble from July 2011 to December 2019

Exclusion Criteria:

* Opposition from patient or parents to participate
* Children who did not effectively suffered a supracondylar humeral fracture

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children operated for a supracondylar humeral fracture in university hospital of Grenoble from July 2011 to December 2019
Sampling Method: Non-Probability Sample
Enrollment: 634 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
functional outcome after supracondylar humeral fracture | 1 day
  Pediatric-Adolescent Shoulder and Elbow Survey (PEDI ASES), rate from 0 to 84, 0 is poor and 84 is excellent
functional outcome after supracondylar humeral fracture | 1 day
  FLYNN'S CRITERIA
functional outcome after supracondylar humeral fracture | 1 day
  range of motion mesured in degrees

SECONDARY OUTCOMES:
post operative complication | 1 day
  identify number and type of complication
time before return to sport | 1 day
  time in days before return to sport
aesthetical prejudice | 1 day
  The Patient and Observer Scar Assement Scale (POSAS), rate from 7 to 70, 7 is excellent and 70 is poor